CLINICAL TRIAL: NCT06004518
Title: The Effect of Sexual Counseling With the PLISSIT Model on Sexual Function and Sexual Quality of Life in Women With Multiple Sclerosis: A Randomized Controlled Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Merve Tuncer, Assist. Prof., Istanbul University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2023/870
Record Dates: First submitted 2023-08-16; First posted 2023-08-22 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Multiple Sclerosis; Female Sexual Dysfunction
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: It was planned in a randomized controlled type.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sexual counselling group (Experimental): Women with MS who are given sexual counseling along with the training booklet will form the sexual counseling group.
  Interventions: Other: sexual counselling with PLISSIT model
- control group (No Intervention): Women with MS who are not given sexual counseling will form the control group.

INTERVENTIONS:
Other: sexual counselling with PLISSIT model — sexual counselling with PLISSIT model
  Arms: sexual counselling group

SUMMARY:
Multiple Sclerosis (MS) is a chronic neuroinflammatory disease of the central nervous system that is common in young ages and women. Plaques formed in MS can develop at any point in the brain and spinal cord, causing various symptoms and adversely affecting the patient's quality of life. Although not counted among the affected neurological systems, one of the most important symptoms experienced by MS patients is sexual dysfunction. Sexual dysfunction in MS may occur due to symptoms of MS such as spasticity, fatigue, and bladder problems, due to the presence of lesions affecting the neural pathways. The most common method used in the treatment of sexual dysfunction in women with MS is sexual counseling. The PLISSIT model is one of the most frequently used models by health professionals in sexual counseling and evaluation. PLISSIT stands for Permission, limited Information, Specific Suggestion and Intensive Therapy.

In this randomized controlled study, the long-term effect of sexual counseling given to female MS patients with the PLISSIT model on sexual function and sexual quality of life will be evaluated. The study is planned to be carried out between July 2023 and December 2024 in the MS and Demyenizing Diseases Unit of Istanbul University Istanbul Medical Faculty Hospital, Department of Neurology. The sample size was calculated as 86, 43 in the sexual counseling group and 43 in the control group, in the G*Power (v3.1.9.7) program using the power analysis method. The data of the study will be collected with the "Descriptive Information Form", "Multiple Sclerosis Intimacy and Sexuality Questionnaire-15", "Sexual Quality of Life Questionnaire for Women", "Patient Health Questionnaire-4" and "Fatigue Severity Scale" developed by the researchers.

The data will be analyzed in SPPS 28 package program. Number, percentage, mean, standard deviation, median and minimum-maximum values will be given in descriptive statistics. The t-test for independent samples/Mann-Whitney U test will be used to compare the mean score of the dependent variables of the two groups. Paired groups t-test/Wilcoxon test will be used in the comparison of each group within the group.

As a result of the research, it is possible to develop an alternative solution approach to the treatment of sexual problems of women with MS by comprehensively evaluating women with MS with sexual problems in line with the PLISSIT model, suggesting solutions, examining the long-term effectiveness of sexual counseling and evaluating the results with concrete, valid and reliable tools. will be provided.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is a chronic autoimmune, inflammatory, demyelinating and/or neurodegenerative disease of the central nervous system. Plaques seen in patients with MS can lead to various symptoms (1). Sexual dysfunction, one of these symptoms, is common in MS patients and negatively affects their quality of life. Sexual dysfunction in MS can be classified as primary, secondary and tertiary. Primary sexual dysfunction is due to the effects of demyelinating lesions on the spinal cord or brain. Secondary dysfunction is due to the physical disorders associated with MS and the side effects of drugs. They indirectly affect the sexual response. Fatigue, loss of attention and concentration, difficulties with movement, coordination disorders, muscle stiffness, bladder and bowel dysfunction, muscle weakness, lower extremity weakness, tremor, pain and drug side effects can be counted as examples of these side effects. Tertiary sexual disorder is the cultural, social and psychological effects of MS. Although sexual dysfunction is a common problem in MS, it is difficult to diagnose and treat because it is not mentioned or questioned. There is no reliable specific treatment for sexual dysfunction for women with MS, but a multidisciplinary approach involving physicians, nurses, sexual therapists, and psychologists is one of the most important components of care for MS patients. It is necessary to provide enough information to the patients about sexual dysfunctions and to enable them to learn the effect of MS on sexuality and current practices in a clear and easy way (3,4).

It is recommended that health professionals use models in order to comprehensively evaluate sexuality and focus on solving sexual problems (5,6). The use of models in the evaluation of sexuality guides health professionals in facilitating the history-taking process and determining sexual problems. The P-LISS-IT model, one of the recommended models for sexual counseling, provides four levels of approach to each problem of the individual: P (Permission): Allowing, Ll (Limited Information): Giving limited information, SS (Specific Suggestions): Giving specific suggestions, IT (Intensive Therapy) is expressed as Intensive Therapy (6). Although there are a limited number of studies showing that sexual counseling based on the PLISSIT model is effective in solving sexual problems in patients with MS, uncertainty about the long-term effects of sexual counseling continues (7-10). In this study, an alternative to the treatment of sexual problems of women with MS was investigated by comprehensively evaluating women with MS with sexual problems in a randomized controlled design in line with the PLISSIT model, examining the long-term effectiveness of sexual counseling by comparing it with the control group, and evaluating the results with concrete, valid and reliable tools. an opportunity to develop a solution approach will be provided. In addition, due to the limited number of studies, it is thought that it will make an important contribution to the literature.

In this study, the following hypotheses will be tested;

1. Sexual functions of women with MS given sexual counseling based on the PLISSIT model are better than women in the control group.
2. Sexual life quality of women with MS who received sexual counseling based on the PLISSIT model is better than women in the control group.

ELIGIBILITY:
Inclusion Criteria:

* • Women between the ages of 18-45,

  * MS diagnosis is finalized,
  * Able to communicate (speak and understand Turkish, no speech disorder),
  * Have not had an attack for at least a month,
  * Expanded Disability Status Scale (EDSS) score of 5.5 or less
  * Those who score 3 or more on each item of the Multiple Sclerosis Intimacy and Sexuality Scale-15
  * Depression and anxiety scores of 3 and below according to the Patient Health Questionnaire-4
  * Those who have a Fatigue Severity Scale score of 8 and below
  * Does not have any additional chronic disease
  * Having a sexual partner and
  * Patients willing to participate in the study will be included in the study.

Exclusion Criteria:

* Women with urinary and stool incontinence problems, menopausal or premenopausal symptoms, a major psychiatric problem and using antidepressant medication, an inflammatory disease such as ankylosing spondylitis or rheumatoid arthritis, substance abuse and those who do not volunteer to participate in the study will not be included.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — female
Enrollment: 86 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
sexual function | 1 year
  Multiple Sclerosis Intimacy and Sexuality Questionnaire

SECONDARY OUTCOMES:
sexual quality of life | 1 year
  Sexual Quality of Life Questionnaire-Female

CONTACTS AND LOCATIONS:
Locations (1):
- Merve TUNCER, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
undecided